CLINICAL TRIAL: NCT04938570
Title: Wearables in Rugby Union: A Protocol for Multimodal Digital Sports-related Concussion Assessment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Northumbria University (Other)
Responsible Party: Sponsor
Other Study IDs: RBHS_01
Record Dates: First submitted 2021-05-18; First posted 2021-06-24 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Concussion, Brain; Sports Injury
MeSH Terms: conditions — Brain Concussion; Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- University-level and amateur rugby players: University-level and amateur rugby players will be recruited and assessed (motor, visual and symptom assessment) over one season ( June 2021 to August 2022).
  Participants will be stratified according to gender (males n≈100, and females n≈100). Although the number of SRC that will be observed during the season is not known, the investigators will compare a number of head injuries/SRC to the results from cohort baseline testing. Participants that do not sustain a concussion will also have follow up testing at the end of the season.

SUMMARY:
The investigators aim to use a repeated measures observational study utilising a battery of multimodal assessment tools (symptom, cognitive, visual, motor). The investigators aim to recruit 200 rugby players (male and female) from University Rugby Union teams and local amateur rugby clubs in the North East of England. The multimodal battery assessment used in this study will compare metrics between digital methods and against traditional assessment.

DETAILED DESCRIPTION:
Background:

Pragmatic challenges remain in the monitoring and return to play (RTP) decisions following suspected Sports Related Concussion (SRC). Reliance on traditional approaches (pen and paper) means players readiness for RTP is often based on self-reported symptom recognition as a marker for full physiological recovery. Non-digital approaches also limit opportunity for robust data analysis which may hinder understanding of the interconnected nature and relationships in deficit recovery. Digital approaches may provide more objectivity to measure and monitor impairments in SRC. Crucially, there is dearth of protocols for SRC assessment and digital devices have yet to be tested concurrently (multimodal) in SRC rugby union assessment. Here the investigators propose a multimodal protocol for digital assessment in SRC, which could be used to enhance traditional sports concussion assessment approach.

Methods:

The investigators aim to use a repeated measures observational study utilising a battery of multimodal assessment tools (symptom, cognitive, visual, motor). The investigators aim to recruit 200 rugby players (male and female) from University Rugby Union teams and local amateur rugby clubs in the North East of England. The multimodal battery assessment used in this study will compare metrics between digital methods and against traditional assessment.

Conclusion: This paper outlines a protocol for a multimodal approach for the use of digital technologies to augment traditional approaches to SRC, which may better inform RTP in rugby union. Findings may shed light on the new ways of working with digital tools in SRC. Multimodal approaches may enhance understanding of the interconnected nature of impairments and provide scalable, more objective assessment and RTP in SRC.

ELIGIBILITY:
Inclusion Criteria:

* 18 years;

  * Have minimal cognitive impairment, defined as a score between 0 and 8 on the Short Blessed test for cognitive function;
  * English as a first language or fluency.
  * Those that have an mTBI/Concussion during the season must have a diagnosis of mTBI from a healthcare professional (physiotherapist or medic) based upon standard criteria or identified head injury from contact sport.

Exclusion Criteria:

* Medical history of a neurological illness that could grossly affect balance or coordination (such as. stroke, greater than mild TBI, lower-extremity amputation, recent lower extremity or spine orthopaedic injury requiring a profile).
* Be a pregnant female
* Have past history of peripheral vestibular pathology or eye movement deficits.
* Be unable to abstain from medication/alcohol 24 hours in advance of testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: University-level and amateur rugby players (males n≈100, and females n≈100) will be recruited and assessed over one season (June 2021 to August 2022). Participants will be stratified according to gender (males and females). Although the number of SRC that will be observed during the season is not known, investigators will compare number of head injuries/SRC to results from cohort baseline testing. Participants that do not sustain a concussion will also have follow up testing at the end of the season
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Step time (mean ± standard deviation) | Participants diagnosed with SRC will be asked to attend a laboratory session/free living assessment at the following subsequent time frames post injury; within 72 hours post, 7-14 days post, within 30 days and 3-6 months
  Altered free-living, quality-based gait/walking patterns measured by digital intertial wearable
Stance time (seconds, mean ± standard deviation) | Participants diagnosed with SRC will be asked to attend a laboratory session/free living assessment at the following subsequent time frames post injury; within 72 hours post, 7-14 days post, within 30 days and 3-6 months
  Altered free-living, quality-based gait/walking patterns measured by digital intertial wearable
Stride time (seconds, mean ± standard deviation) | Participants diagnosed with SRC will be asked to attend a laboratory session/free living assessment at the following subsequent time frames post injury; within 72 hours post, 7-14 days post, within 30 days and 3-6 months
  Altered free-living, quality-based gait/walking patterns measured by digital intertial wearable
Swing time (seconds, mean ± standard deviation) | Participants diagnosed with SRC will be asked to attend a laboratory session/free living assessment at the following subsequent time frames post injury; within 72 hours post, 7-14 days post, within 30 days and 3-6 months
  Altered free-living, quality-based gait/walking patterns measured by digital intertial wearable
Stride length (cm, mean ± standard deviation) | Participants diagnosed with SRC will be asked to attend a laboratory session/free living assessment at the following subsequent time frames post injury; within 72 hours post, 7-14 days post, within 30 days and 3-6 months
  Altered free-living, quality-based gait/walking patterns measured by digital intertial wearable
Stride velocity (cms-1), mean ± standard deviation) | Participants diagnosed with SRC will be asked to attend a laboratory session/free living assessment at the following subsequent time frames post injury; within 72 hours post, 7-14 days post, within 30 days and 3-6 months
  Altered free-living, quality-based gait/walking patterns measured by digital intertial wearable

SECONDARY OUTCOMES:
Number of turns per hour (n, mean ± standard deviation) | Participants diagnosed with SRC will be asked to attend a laboratory session/free living assessment at the following subsequent time frames post injury; within 72 hours post, 7-14 days post, within 30 days and 3-6 months
  Altered free-living, quality-based turning patterns measured by digital intertial wearable
Turn angle (°, mean ± standard deviation) | Participants diagnosed with SRC will be asked to attend a laboratory session/free living assessment at the following subsequent time frames post injury; within 72 hours post, 7-14 days post, within 30 days and 3-6 months
  Altered free-living, quality-based turning patterns measured by digital intertial wearable
Turn duration (seconds, mean ± standard deviation)) | Participants diagnosed with SRC will be asked to attend a laboratory session/free living assessment at the following subsequent time frames post injury; within 72 hours post, 7-14 days post, within 30 days and 3-6 months
  Altered free-living, quality-based turning patterns measured by digital intertial wearable
Turn velocity (°/seconds, mean ± standard deviation)) | Participants diagnosed with SRC will be asked to attend a laboratory session/free living assessment at the following subsequent time frames post injury; within 72 hours post, 7-14 days post, within 30 days and 3-6 months
  Altered free-living, quality-based turning patterns measured by digital intertial wearable

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Powell D, Stuart S, Godfrey A. Wearables in rugby union: A protocol for multimodal digital sports-related concussion assessment. PLoS One. 2021 Dec 22;16(12):e0261616. doi: 10.1371/journal.pone.0261616. eCollection 2021. PMID 34936689

DOCUMENTS (1):
  • Informed Consent Form (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT04938570/ICF_000.pdf